CLINICAL TRIAL: NCT02489422
Title: GI 1549: PROGRAMS TO SUPPORT YOU DURING CHEMOTHERAPY (PRO-YOU) A Randomized Controlled Pilot Study of Yoga Compared to an Attention Control in Patients Receiving Chemotherapy
Brief Title: Programs To Support You During Chemotherapy
Acronym: PRO-YOU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00038321; NCI-2015-01042 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 01716 (Other: Comprehensive Cancer Center of Wake Forest University); K01AT008219 (NIH); P30CA068485 (NIH)
Record Dates: First submitted 2015-06-29; First posted 2015-07-03 (Estimated); Results first posted 2021-05-27 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-09

CONDITIONS: Depression; Fatigue; Stage IIA Colorectal Cancer; Stage IIB Colorectal Cancer; Stage IIC Colorectal Cancer; Stage IIIA Colorectal Cancer; Stage IIIB Colorectal Cancer; Stage IIIC Colorectal Cancer; Stage IVA Colorectal Cancer; Stage IVB Colorectal Cancer; Pancreatic Cancer; Esophageal Cancer; Appendix Cancer; Stomach Cancer; Gallbladder Cancer; Liver Cancer; Small Intestine Cancer; Large Intestine Cancer; Anal Cancer; Biliary Tract Cancer; Gastrointestinal Stromal Cancer
MeSH Terms: conditions — Depression; Fatigue; Colorectal Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms; Appendiceal Neoplasms; Stomach Neoplasms; Gallbladder Neoplasms; Liver Neoplasms; Colonic Neoplasms; Anus Neoplasms; Biliary Tract Neoplasms | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Yoga Skills Training) (Experimental): Patients participate in YST consisting of four 30 minute in-person yoga sessions at weeks 2, 4, 6, and 8 that instructs skills to enhance mindfulness and promote relaxation, through instruction of awareness, movement, breathing practices, and meditation.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Other: Daily Survey Administration; Behavioral: Yoga Skills Training; Other: Actigraphy Assessment
- Group II (Attention Control) (Active Comparator): Patients participate in four 30 minute in-person sessions of supportive conversation at weeks 2, 4, 6, 8.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Other: Daily Survey Administration; Behavioral: Attention Control; Other: Actigraphy Assessment

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies
Other: Daily Survey Administration — Ancillary studies
Behavioral: Yoga Skills Training — The YST intervention consists of four 30 minute in-person sessions that instructs skills to enhance mindfulness and promote relaxation. Participants will also be encouraged to practice daily at home.
  Other Names: yoga; YST
  Arms: Group I (Yoga Skills Training)
Behavioral: Attention Control — The AC intervention consists of four 30 minute in-person sessions of supportive conversation. In addition, the interventionist will recommend that the patients write brief diary entries daily at home.
  Other Names: empathic attention control; supportive conversation; caring attention control
  Arms: Group II (Attention Control)
Other: Actigraphy Assessment — Ancillary studies
  Other Names: Circadian Disruption - daily

SUMMARY:
This randomized pilot trial studies how well two supportive programs work for improving fatigue and depressive symptoms in patients with GI undergoing chemotherapy. Possible mediators such as psychological stress, circadian disruption, and inflammation, will also be explored.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To conduct a pilot randomized controlled trial of the yoga skills training (YST) versus a caring attention control (AC) group among adults with colorectal cancer (CRC) receiving chemotherapy to determine preliminary efficacy for the primary outcome of fatigue, secondary outcome of depressive symptoms, and possible mediators (i.e., psychological stress, circadian disruption, inflammation) as assessed by standard measures.

SECONDARY OBJECTIVES:

I. To measure the impact of the YST versus the AC on daily assessments of fatigue, depressive symptoms, and proposed mediators in the same trial and explore relationships among daily and standard assessments.

II. To qualitatively assess perceived efficacy of the YST and AC and acceptability of new methodology through semi-structured interviews in a subset of 20-40 participants.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (YST): Patients participate in YST consisting of four 30 minute in-person yoga sessions at weeks 2, 4, 6, and 8 that instructs skills to enhance mindfulness and promote relaxation, through instruction of awareness, movement, breathing practices, and meditation.

GROUP II (AC): Patients participate in four 30 minute in-person sessions of supportive conversation at weeks 2, 4, 6, and 8.

After completion of study, patients are followed up at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to receive first-line Fluorouracil (5FU)-based intravenous chemotherapy treatment for a gastrointestinal cancer (stages II-IV)
* Have an Eastern Cooperative Oncology Group performance status of =< 1
* Ability to understand and the willingness to sign and informed consent document in English

Exclusion Criteria:

* Has a self-reported history of diagnosed uncontrolled obstructive sleep apnea (ok if using CPAP), sleep-related seizures, sleep walking more than one time per week, restless leg syndrome, or a job with night shifts

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-08; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sohl, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (2):
- United States (2):
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Started | 23 | 21
Completed | 23 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control) | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (11.3) | 56.0 (12.0) | 58.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 23 | 20 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 20 | 18 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS)
Description: Fatigue will be assessed with the 7-item measure of Fatigue from the PROMIS-cancer specifically designed for use in cancer patients. These tests will be evaluated using mixed-effects (or multilevel) generalized linear modeling procedures. Score range 1 - never, 2 - rarely, 3 - sometimes, 4 - often and 5 - always. Total scores can range from 24 to 86, with higher scores indicating greater fatigue.
Time Frame: At baseline, 8 weeks, 10 weeks and 14 weeks after start of intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 23 | 21
score on a scale
  Baseline | 53.1 (1.8) | 56.8 (1.9)
  8 weeks | 53.0 (2.1) | 57.2 (2.2)
  10 weeks | 51.1 (2.2) | 57.2 (2.4)
  14 weeks | 55.4 (2.2) | 60.6 (2.3)

2. Secondary Outcome: Circadian Disruption (Daily)
Description: Circadian disruption will be assessed with actigraphy. Circadian disruption is defined as a ratio of nighttime activity to daytime activity with higher scores indicating greater circadian disruptions. Summaries of the proportion and frequency of missing daily assessments will inform the feasibility of collecting this type of data.
Time Frame: At 0-2 weeks after start of intervention
Population: Participants analyzed represents the number of participants that completed the analysis and had data for this outcome measure out of the total number of participants for the trial.
Measure: Mean (Standard Error); unit: days
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 23 | 21
days | 11.5 (2.8) | 9.9 (3.4)

3. Secondary Outcome: Circadian Disruption (Daily)
Description: as for outcome 2
Time Frame: At 8-10 weeks after start of intervention
Population: The number of participants is the actual number that completed this portion of the outcome measure during this timeframe that had measurable data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 21 | 19
days | 11.8 (2.3) | 11.9 (2.3)

4. Secondary Outcome: Circadian Disruption (Recalled)
Description: Circadian disruption will be assessed with measures of activity and rest. Activity will be measured using the 3-item Godin's leisure score index (LSI), previously used with colorectal cancer patients during chemotherapy. Rest will be assessed with the 8-item PROMIS sleep disturbance short-form. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
Time Frame: At baseline, 8 weeks, 10 weeks and 14 weeks after start of intervention
Population: Numbers may vary based on number of participants that actually completed intervention materials
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 23 | 21
score on a scale
  Baseline leisure score index (LSI): number analyzed (Participants) | 21 | 17
  Baseline leisure score index (LSI) | 19.6 (5.4) | 19.9 (3.6)
  8 weeks leisure score index (LSI): number analyzed (Participants) | 15 | 16
  8 weeks leisure score index (LSI) | 24.1 (7.1) | 23.9 (6.2)
  10 weeks leisure score index (LSI): number analyzed (Participants) | 20 | 13
  10 weeks leisure score index (LSI) | 19.8 (4.4) | 29.7 (12.0)
  14 weeks leisure score index: number analyzed (Participants) | 16 | 13
  14 weeks leisure score index | 24.1 (5.5) | 38.1 (12.8)

5. Secondary Outcome: Depressive Symptoms Assessed by PROMIS
Description: Will be assessed with the standardized 10-item PROMIS-cancer depressive symptoms short-form. These tests will be evaluated using mixed-effects (or multilevel) generalized linear modeling procedures. Scoring scale range from 1 - never, 2 - rarely, 3 - sometimes, 4 - often and 5 - always. The higher the score the more depressive the symptoms. Scores on the short form range from 10 to 81.3; 10-55 is "normal", 55.1-59.9 "mild", 60-64.25 "moderate", and over 64.26 "severe" depression.
Time Frame: At baseline, 8 weeks, 10 weeks and 14 weeks after start of intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 23 | 21
score on a scale
  Baseline | 49.9 (1.9) | 51.4 (2.0)
  8 weeks | 47.4 (2.0) | 51.2 (2.1)
  10 weeks | 46.6 (2.3) | 50.5 (2.5)
  14 weeks | 49.1 (2.0) | 50.2 (2.1)

6. Secondary Outcome: Fatigue (Daily)
Description: Fatigue will be assessed with 3 items selected from the PROMIS measure of fatigue validated for use in daily diaries. Scoring scale range from 1 - never, 2 - rarely, 3 - sometimes, 4 - often and 5 - always. The higher the score the more fatigued the participants. Scores on the short form range from 0 to 81.3; 0-55 is "normal", 55.1-59.9 "mild", 60-64.25 "moderate", and over 64.26 "severe" fatigue.
Time Frame: At 0-2 weeks and 8-10 weeks after start of intervention
Population: Numbers may vary based on number of participants that actually completed intervention materials
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 23 | 21
score on a scale
  0-2 weeks: number analyzed (Participants) | 23 | 19
  0-2 weeks | 49.18 (1.73) | 53.27 (1.92)
  8-10 weeks: number analyzed (Participants) | 16 | 14
  8-10 weeks | 51.00 (2.06) | 53.29 (2.38)

7. Secondary Outcome: Depressive Symptoms (Daily)
Description: Depressive symptoms will be assessed with 3 items selected from the PROMIS measure of depression validated for use in daily diaries. Scoring scale range from 1 - never, 2 - rarely, 3 - sometimes, 4 - often and 5 - always. The higher the score the more depressive symptoms the participants exhibited. scores on the short form range from 0 to 81.3; 0-55 is "normal", 55.1-59.9 "mild", 60-64.25 "moderate", and over 64.26 "severe" depression.
Time Frame: At 0-2 weeks and 8-10 weeks after start of intervention
Population: Numbers may vary based on number of participants that actually completed intervention materials
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 23 | 21
score on a scale
  0-2 weeks: number analyzed (Participants) | 20 | 19
  0-2 weeks | 43.96 (1.52) | 45.49 (1.82)
  8-10 weeks: number analyzed (Participants) | 16 | 14
  8-10 weeks | 44.38 (2.36) | 44.58 (1.89)

8. Secondary Outcome: Interleukin 6 [IL-6] Measured Using High-sensitivity Quantikine Immunoassay Kits
Description: Inflammatory cytokines (i.e., interleukin 6 [IL-6], soluble tumor necrosis factor receptor 1 [sTNF-R1], and tumor necrosis factor alpha [TNF-alpha]) that have been associated with fatigue during treatment for gastrointestinal cancer and influenced by yoga practice will be measured using high-sensitivity Quantikine immunoassay kits.
Time Frame: At 2 weeks after start of intervention
Population: The number of participants represents the number that completed data to be analyzed for this particular outcome measure.
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 16 | 13
pg/ml | 5.6 [3.4 to 9.2] | 4.6 [2.8 to 7.8]

9. Secondary Outcome: Interleukin 6 [IL-6] Measured Using High-sensitivity Quantikine Immunoassay Kits
Description: Inflammatory cytokines (i.e., interleukin 6 [IL-6], soluble tumor necrosis factor receptor 1 [sTNF-R1], and tumor necrosis factor alpha [TNF-alpha]) that have been associated with fatigue during treatment for gastrointestinal cancer and influenced by yoga practice will be measured using high-sensitivity Quantikine immunoassay kits. ). All samples will be assayed in duplicate and the average of the two measures will be used for data analyses.
Time Frame: At 10 weeks after start of intervention
Population: The number of participants represents the number that completed data to be analyzed for this particular outcome measure.
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 16 | 13
pg/ml | 0.58 [0.38 to 0.90] | 0.58 [0.38 to 0.90]

10. Secondary Outcome: Soluble Tumor Necrosis Factor Receptor 1 [sTNF-R1] Measured Using High-sensitivity Quantikine Immunoassay Kits
Description: as for outcome 8
Time Frame: At 2 weeks after start of intervention
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 16 | 13
pg/ml | 1633.8 [1222.1 to 2184.1] | 1727.5 [1281.6 to 2328.6]

11. Secondary Outcome: Soluble Tumor Necrosis Factor Receptor 1 [sTNF-R1] Measured Using High-sensitivity Quantikine Immunoassay Kits
Description: Inflammatory cytokines (i.e., interleukin 6 [IL-6], soluble tumor necrosis factor receptor 1 [sTNF-R1], and tumor necrosis factor alpha [TNF-alpha]) that have been associated with fatigue during treatment for gastrointestinal cancer and influenced by yoga practice will be measured using high-sensitivity Quantikine immunoassay kits. All samples will be assayed in duplicate and the average of the two measures will be used for data analyses.
Time Frame: At 10 weeks after start of intervention
Population: The number of participants represents the number that completed data to be analyzed for this particular outcome measure.
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 16 | 13
pg/ml | 0.87 [0.78 to 0.97] | 0.87 [0.78 to 0.97]

12. Secondary Outcome: Tumor Necrosis Factor Alpha [TNF-alpha] Measured Using High-sensitivity Quantikine Immunoassay Kits
Description: as for outcome 8
Time Frame: At 2 weeks after start of intervention
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 16 | 13
pg/ml | 1.6 [1.1 to 2.1] | 1.7 [1.2 to 2.3]

13. Secondary Outcome: Tumor Necrosis Factor Alpha [TNF-alpha] Measured Using High-sensitivity Quantikine Immunoassay Kits
Description: as for outcome 11
Time Frame: At 10 weeks after start of intervention
Population: Numbers may vary based on number of participants that actually completed intervention materials
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 16 | 13
pg/ml | 1.01 [0.91 to 1.13] | 1.01 [0.91 to 1.13]

14. Secondary Outcome: Psychological Stress Assessed by the Perceived Stress Scale (PSS)
Description: Psychological stress will be assessed by the 10-item PSS. The PSS has 2 factors (stress and counter stress). Scoring scale range from 0 - never, 1 - almost never, 2 - sometimes, 3 - fairly often and 4 - very often. Score range is 0-40. A higher score represents more of the concept being measured.
Time Frame: At baseline, 8 weeks, 10 weeks and 14 weeks after start of intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 22 | 20
score on a scale
  Baseline, mean | 14.7 (1.5) | 16.5 (1.6)
  8 weeks | 11.4 (1.8) | 13.7 (1.9)
  10 weeks | 12.1 (1.8) | 12.3 (2.1)
  14 weeks | 12.5 (1.8) | 13.6 (1.9)

15. Secondary Outcome: Psychological Stress Assessed by the PSS (Daily)
Description: Psychological stress will be assessed daily with two items from the 4-item PSS that would be on the same factor to optimize internal consistency. Scoring scale range from 1 - never, 2 - rarely, 3 - sometimes, 4 - often and 5 - always. A mean of the participants scores was taken.
Time Frame: At 0-2 weeks and 8-10 weeks after start of intervention
Population: Numbers may vary based on number of participants that actually completed intervention materials
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 20 | 19
score on a scale
  0-2 weeks, mean | 1.34 (0.36) | 1.58 (0.42)
  8-10 weeks, mean: number analyzed (Participants) | 16 | 14
  8-10 weeks, mean | 1.69 (0.55) | 1.78 (0.45)

16. Secondary Outcome: Regulation of Psychological Stress Assessed by the Positive and Negative Affect Schedule-Expanded Form (Daily)
Description: Regulation of psychological stress will be assessed daily with the 3-item serenity subscale (calm, relaxed, at ease) from the Positive and Negative Affect Schedule-Expanded Form. Each item is rated on a five-point Likert Scale, ranging from 1 = Very Slightly or Not at all to 5 = Extremely. Positive Affect Score: Scores can range from 10 - 50, with higher scores representing higher levels of positive affect and lower scores representing lower levels of negative affect.
Time Frame: At 0-2 weeks and 8-10 weeks after start of intervention
Population: Numbers may vary based on number of participants that actually completed intervention materials
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 20 | 19
score on a scale
  0-2 weeks, mean | 10.51 (0.55) | 9.59 (0.66)
  8-10 weeks, mean: number analyzed (Participants) | 16 | 14
  8-10 weeks, mean | 10.53 (0.74) | 10.36 (0.84)

17. Secondary Outcome: Regulation of Psychological Stress Assessed Using the Cancer Behavior Inventory
Description: Regulation of psychological stress will be determined by ratings on four of the seven factors of the Cancer Behavior Inventory, which assess self-efficacy for stress management, coping with treatment-related side-effects, accepting cancer/maintaining positive attitude, and affective regulation. Scale ranged from 1-9 (1 - 3 not at all confident; 4-6 moderately confident and 7-9 totally confident). 4 of the 7 items from the Cancer Behavior Inventory (V2.0) were used with each item's score ranges from 0-50 with higher scores indicating more confidence in the item.
Time Frame: At baseline, 8 weeks, 10 weeks and 14 weeks after start of intervention
Population: Numbers may vary based on number of participants that actually completed intervention materials
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 23 | 20
score on a scale
  Baseline - Stress management | 34.8 (1.4) | 34.2 (1.5)
  Baseline - Coping with treatment-related side effects: number analyzed (Participants) | 22 | 20
  Baseline - Coping with treatment-related side effects | 33.1 (1.8) | 30.6 (1.8)
  Baseline - Accepting cancer/maintaining positive attitude | 37.8 (1.3) | 39.3 (0.9)
  Baseline - Affective regulation: number analyzed (Participants) | 22 | 20
  Baseline - Affective regulation | 28.2 (1.6) | 29.9 (1.6)
  8 weeks - Stress management: number analyzed (Participants) | 18 | 16
  8 weeks - Stress management | 38.1 (1.3) | 38.6 (1.9)
  8 weeks - Coping with treatment-related side effects: number analyzed (Participants) | 18 | 16
  8 weeks - Coping with treatment-related side effects | 37.1 (1.7) | 35.4 (2.1)
  8 weeks - Accepting cancer/maintaining positive attitude: number analyzed (Participants) | 18 | 16
  8 weeks - Accepting cancer/maintaining positive attitude | 40.4 (1.2) | 38.9 (1.6)
  8 weeks - Affective regulation: number analyzed (Participants) | 18 | 16
  8 weeks - Affective regulation | 29.8 (2.1) | 31.8 (2.1)
  10 weeks - Stress management: number analyzed (Participants) | 20 | 13
  10 weeks - Stress management | 38.2 (1.1) | 38.5 (1.6)
  10 weeks - Coping with treatment-related side effects: number analyzed (Participants) | 20 | 13
  10 weeks - Coping with treatment-related side effects | 36.8 (1.6) | 37.5 (2.3)
  10 weeks - Accepting cancer/maintaining positive attitude: number analyzed (Participants) | 20 | 13
  10 weeks - Accepting cancer/maintaining positive attitude | 40.6 (0.9) | 40.6 (1.6)
  10 weeks - Affective regulation: number analyzed (Participants) | 20 | 13
  10 weeks - Affective regulation | 30.1 (2.2) | 33.1 (2.3)
  14 weeks - Stress management: number analyzed (Participants) | 17 | 15
  14 weeks - Stress management | 39.2 (1.4) | 40.1 (1.1)
  14 weeks - Coping with treatment-related side effects: number analyzed (Participants) | 17 | 15
  14 weeks - Coping with treatment-related side effects | 37.0 (1.7) | 38.4 (1.5)
  14 weeks - Accepting cancer/maintaining positive attitude: number analyzed (Participants) | 17 | 15
  14 weeks - Accepting cancer/maintaining positive attitude | 40.0 (1.2) | 41.1 (1.0)
  14 weeks - Affective regulation: number analyzed (Participants) | 17 | 15
  14 weeks - Affective regulation | 32.3 (2.1) | 34.0 (1.9)

18. Secondary Outcome: Minutes of Home Practice Completed
Description: Participants will keep daily paper logs of their home practice. In addition, one item will ask via the daily automated survey how many minutes participants practiced the intervention that day for two weeks after completion of the intervention.
Time Frame: Up 10 weeks after start of intervention
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 16 | 14
minutes | 11.2 (1.9) | 12.1 (6.3)

19. Secondary Outcome: Percent of Planned In Person Intervention Sessions Attended
Description: Percent of all assessments completed and timeliness of completion will be tracked.
Time Frame: At baseline, 2 weeks, 8 weeks, 10 weeks and 14 weeks after start of intervention
Population: Four in-person interventions were performed per participant at weeks 2, 4, 6, and 8. A total of 92 interventions were available for completion for Group I. A total of 84 interventions were available for completion for Group II.
Measure: Number; unit: total interventions actually completed
Units Other Than Participants: total of interventions available
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
Number analyzed (Participants) | 23 | 21
Number analyzed (total of interventions available) | 92 | 84
total interventions actually completed | 68 | 72

20. Secondary Outcome: Number of Participants With Successful Qualitative Data Collection
Description: Qualitative feedback will be assessed with a semi-structured interview conducted after completion of all assessments. Qualitative information gained will enrich quantitative results and inform the protocol of a larger trial.
Time Frame: At 14 weeks after start of intervention
Population: As per the protocol, this outcome was intended to be combined after all other data collection is complete to solicit feedback as a group on the acceptability of data collection methods, the participants' experience with both the interventions (e.g., expected efficacy, what was useful), and barriers and facilitators to home practice. It was not intended to be separated but as overall feedback.
Measure: Count of Participants; unit: Participants
Groups:
- Qualitative Interviews - Combined: Qualitative feedback will be assessed with a semi-structured interview conducted after completion of all assessments.
Arm/Group | Qualitative Interviews - Combined
Number analyzed (Participants) | 43
Participants | 30

ADVERSE EVENTS:
Time Frame: Over 8 weeks
Arm/Group | Group I (Yoga Skills Training) | Group II (Attention Control)
All-Cause Mortality (participants affected / at risk) | 2/23 | 2/21
Serious Adverse Events (participants affected / at risk) | 4/23 | 3/21
Other Adverse Events (participants affected / at risk) | 1/23 | 2/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Yoga Skills Training) (N=23) | Group II (Attention Control) (N=21)
Death (General disorders) | 2 (2) | 2 (2)
Bowel perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Yoga Skills Training) (N=23) | Group II (Attention Control) (N=21)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT02489422/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT02489422/ICF_001.pdf